CLINICAL TRIAL: NCT03469622
Title: EndoRings Versus Standard Colonoscopy for Adenoma Detection
Brief Title: EndoRings Colonoscopy for Adenoma Detection
Acronym: ER
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Helios Albert-Schweitzer-Klinik Northeim (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Factorial | Masking: Single | Purpose: Diagnostic
Other Study IDs: HRC 047721
Record Dates: First submitted 2018-03-06; First posted 2018-03-19 (Actual); Last update posted 2019-02-12 (Actual); Status verified 2019-02

CONDITIONS: Adenoma
Keywords: Adenoma; Polyp; EndoRings; Colonoscopy; Endoscopic device; Colon cancer screening
MeSH Terms: conditions — Adenoma; Polyps

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- EndoRings (Active Comparator): Colonoscopy is performed with the EndoRings attached
  Interventions: Device: EndoRings
- Standard Colonoscopy (Active Comparator): Standard colonoscopy without any additional devices
  Interventions: Device: Standard colonoscopy

INTERVENTIONS:
Device: EndoRings — EndoRings-assisted colonoscopy
  Arms: EndoRings
Device: Standard colonoscopy — Standard colonoscopy without any additional devices
  Arms: Standard Colonoscopy

SUMMARY:
Adenoma detection rate (ADR) in colon cancer screening is most important for avoiding colon cancer development. Recent studies suggest a benefit of endoscopic devices attached to the distal tip of the colonoscope for improving the ADR. This work is the first GERMAN randomized controlled trial comparing standard colonoscopy with EndoRIngs-assisted colonoscopy.

EndoRings is a new FDA approved device that is attached to the distal tip of the colonoscope. Better Polyp detection is suspected by flattening the mucosal folds during withdrawal

ELIGIBILITY:
Inclusion Criteria:

* indication for colonoscopy (screening, surveillance, diagnostic)
* age ≥ 45 years
* ability to give informed consent

Exclusion Criteria:

* pregnancy
* age <45 years
* known colonic strictures
* chronic inflammatory bowel disease
* active inflammation
* s/p colonic resection
* bleeding disorder

Min Age: 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 225 (Estimated)
Dates: Start 2018-03-27 (Actual); Primary Completion 2019-12-31 (Estimated); Study Completion 2019-12-31 (Estimated)

PRIMARY OUTCOMES:
Adenoma detection rate | during colonoscopy

CONTACTS AND LOCATIONS:
Overall Officials: Tobias Meister, Prof. Dr., Principal Investigator — HELIOS Albert-Schweitzer Klinik; Ralf Kiesslich, Prof. Dr., Principal Investigator — HELIOS HSK Kliniken Wiesbaden
Locations (5):
- Germany (5):
  - HELIOS HSK Kliniken, Wiesbaden, Hesse
  - Department of Gastroenterology, University Medical Center, Göttingen, Lower Saxony
  - HELIOS St. Marienberg Klinik Helmstedt, Helmstedt
  - Helios Albert-Schweitzer-Hospital, Academic University Teaching Hospital, Northeim
  - HELIOS Medical Center Siegburg, Siegburg